CLINICAL TRIAL: NCT04920123
Title: Towards the Development of a Mobile-health Technology Designed to Encourage the Use of Serious Game-based Interventions in Patients With Mild Cognitive Impairment Outside the Clinic
Brief Title: Serious Game-based Interventions in Patients With Mild Cognitive Impairment Outside the Clinic
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Massachusetts, Amherst (Other)
Collaborators: Rutgers, The State University of New Jersey (Other); Université de Montréal (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 2585
Record Dates: First submitted 2021-06-03; First posted 2021-06-09 (Actual); Results first posted 2025-08-07 (Actual); Last update posted 2025-08-07 (Actual); Status verified 2025-06

CONDITIONS: Mild Cognitive Impairment
MeSH Terms: conditions — Cognitive Dysfunction

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Game Intervention (Experimental): Study participants play Neuro-World 30 minutes per day, twice a week for 12 weeks in your home settings (24 times).
  Interventions: Device: Neuro-World
- No Intervention (No Intervention): Study participants do not engage in any cognitive training.

INTERVENTIONS:
Device: Neuro-World — Neuro-World is a collection of six games that are developed for cognitive training that focuses on memory and attention.
  Arms: Game Intervention

SUMMARY:
This study will evaluate the therapeutic efficacy of Neuro-World cognitive training games (Woorisoft, S. Korea) in patients with mild cognitive impairment.

DETAILED DESCRIPTION:
This study will be a cross-over randomized controlled trial.

Fifty participants will be enrolled and randomly assigned to group A or group B.

Group A will self-administer Neuro-World cognitive training games for 30 minutes a day, twice a week for 12 weeks in the home setting (i.e., intervention period). For the following 12 weeks, the participants will not engage in any therapist-supervised cognitive therapies (i.e., no-intervention period).

Group B will not engage in any therapist-supervised cognitive therapies (i.e., no-intervention period). For the following 12 weeks, the participants will self-administer Neuro-World cognitive training games for 30 minutes a day, twice a week in the home setting (i.e., intervention period).

All the participants in both groups will receive phone calls twice a week to 1) provide feedback on their adherence to Neuro-World cognitive training (during the intervention period) and 2) learn any significant changes in the level of their daily activities (during the no-intervention period and the intervention period).

ELIGIBILITY:
Inclusion Criteria:

* Seventeen points or greater and smaller than twenty-six points on the Montreal Cognitive Assessment (MoCA)
* Fifty-five years old and above
* Minimal technological literacy (i.e. ability to use a tablet independently)
* Having a computer for online videoconferencing-based communication (necessary for online cognitive assessments)

Exclusion Criteria:

* Confounding neurological and psychiatric disorders
* History of traumatic brain injury
* Clinically known hearing or vision impairment
* Severe upper-limb motor impairments that could impact the use of mobile devices
* Clinical presentations suggestive of dementia with Lewy bodies, progressive supranuclear palsy, multiple system atrophy, or vascular parkinsonism
* Diagnosis of dementia
* Major depression
* Any significant upper-limb impairment that could affect tablet use
* Participation in any other therapist-supervised cognitive training

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2022-02-17 (Actual); Primary Completion 2025-03-31 (Actual); Study Completion 2025-03-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sunghoon I Lee, PhD, Principal Investigator — University of Massachusetts, Amherst
Locations (2):
- United States (2):
  - University of Massachusetts, Amherst, Amherst, Massachusetts
  - The State University of New Jersey, Rutgers, Newark, New Jersey

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited remotely across the United States and Canada through email, phone, and social media. Of the 155 individuals contacted, 41 were screened for eligibility via videoconference. Fifteen met inclusion criteria and were enrolled in the study. Three participants later discontinued participation.
Pre-assignment Details: Fifteen participants were enrolled and randomized into two groups. Three participants discontinued participation during the study. No significant events such as washout or run-in periods occurred prior to group assignment.
  Four caregivers were enrolled to assist with technical arrangements and help manage study logistics. Two caregivers discontinued participation during the study after the participants they were assisting withdrew.
Groups:
- Group A: Intervention, Then Non-intervention: Group A will self-administer Neuro-World cognitive training games for 30 minutes per day, twice a week, for 12 weeks in a home setting (intervention period). This will be followed by 12 weeks without any therapist-supervised cognitive therapies (non-intervention period).
- Group B: Non-intervention, Then Intervention: Group B will first complete a 12-week non-intervention period without therapist-supervised cognitive therapies. This will be followed by 12 weeks of self-administered Neuro-World cognitive training games for 30 minutes per day, twice a week, in a home setting (intervention period).
- Caregivers: Caregivers are optionally enrolled to assist with technical arrangements and help manage study logistics. No interventions are administered to the caregiver group.
Period: First Intervention (12 Weeks)
Arm/Group | Group A: Intervention, Then Non-intervention | Group B: Non-intervention, Then Intervention | Caregivers
Started | 8 | 7 | 4
Completed | 6 | 6 | 2
Not Completed | 2 | 1 | 2
Not completed — Withdrawal by Subject | 2 | 1 | 2
Period: Second Intervention (12 Weeks)
Arm/Group | Group A: Intervention, Then Non-intervention | Group B: Non-intervention, Then Intervention | Caregivers
Started | 6 | 6 | 2
Completed | 6 | 6 | 2
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group A: Intervention, Then Non-intervention | Group B: Non-intervention, Then Intervention | Caregivers | Total
Number analyzed (Participants) | 8 | 7 | 4 | 19
Age, Continuous [Mean (Standard Deviation); unit: Years] | 63.3 (13.2) | 57.8 (10.1) | 48.0 (19.6) | 62.4 (11.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 5 | 0 | 10
  Male | 3 | 2 | 4 | 9
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 1 | 1
  Not Hispanic or Latino | 6 | 6 | 3 | 15
  Unknown or Not Reported | 2 | 1 | 0 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 2 | 2 | 1 | 5
  White | 5 | 5 | 3 | 13
  More than one race | 1 | 0 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 8 | 7 | 4 | 19

OUTCOME MEASURES:

1. Primary Outcome: Change in Montreal Cognitive Assessment (MoCA)
Description: MoCA scores range between 0 and 30. Higher scores indicate better cognitive function. The change in MoCA scores was measured from baseline to 12 weeks
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Game Intervention | No Intervention
Number analyzed (Participants) | 12 | 12
score on a scale | -2.0 (3.24) | 2.8 (1.88)
Statistical Analysis 1: Comparison: Game Intervention vs No Intervention; Null hypothesis: no improvement or worse with intervention Alternative hypothesis: improvement with intervention; Test type: Superiority; p = 0.997, t-test, 1 sided — The threshold for statistical significance was p=0.05

2. Secondary Outcome: Change in Mini-Mental State Examination (MMSE)
Description: MMSE scores range between 0 and 30. Higher scores indicate better cognitive function. The change in MMSE scores was measured from baseline to 12 weeks
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Game Intervention | No Intervention
Number analyzed (Participants) | 12 | 12
score on a scale | 0.5 (2.14) | 0.5 (1.85)
Statistical Analysis 1: Comparison: Game Intervention vs No Intervention; Null hypothesis: no improvement or worse with intervention Alternative hypothesis: improvement with intervention; Test type: Superiority; p = 0.500, t-test, 1 sided — The threshold for statistical significance was p=0.05

3. Secondary Outcome: Change in Digit Forward Span (DFS)
Description: DFS scores range between 0 and 14. Higher scores indicate better cognitive function. The change in DFS scores was measured from baseline to 12 weeks
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Game Intervention | No Intervention
Number analyzed (Participants) | 12 | 12
score on a scale | -0.2 (1.74) | 0.8 (1.96)
Statistical Analysis 1: Comparison: Game Intervention vs No Intervention; Null hypothesis: no improvement or worse with intervention Alternative hypothesis: improvement with intervention; Test type: Superiority; p = 0.821, t-test, 1 sided — The threshold for statistical significance was p=0.05

4. Secondary Outcome: Change in Digit Backward Span (DBS)
Description: DBS scores range between 0 and 14. Higher scores indicate better cognitive function. The change in DBS scores was measured from baseline to 12 weeks
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Game Intervention | No Intervention
Number analyzed (Participants) | 12 | 12
score on a scale | -1.1 (1.55) | 1.4 (1.50)
Statistical Analysis 1: Comparison: Game Intervention vs No Intervention; Null hypothesis: no improvement or worse with intervention Alternative hypothesis: improvement with intervention; Test type: Superiority; p = 0.995, t-test, 1 sided — The threshold for statistical significance was p=0.05

5. Secondary Outcome: Change in Geriatric Depression Scale (GDS)
Description: GDS scores range between 0 and 15. Higher scores indicate more severe depression. The change in GDS scores was measured from baseline to 12 weeks
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Game Intervention | No Intervention
Number analyzed (Participants) | 12 | 12
score on a scale | -0.8 (1.77) | 0.2 (0.69)
Statistical Analysis 1: Comparison: Game Intervention vs No Intervention; Null hypothesis: no improvement or worse with intervention Alternative hypothesis: improvement with intervention; Test type: Non-Inferiority — Higher scores indicate more severe depression; p = 0.076, t-test, 1 sided

6. Secondary Outcome: Change in Short Form 36 (SF-36) Mental Component Summary Score
Description: SF-36 consists of eight health domains, each scored from 0 to 100, with higher scores indicating more favorable health states. In this study, we report the Mental Component Summary (MCS) score, a norm-based composite score derived from relevant mental health domains. The MCS is standardized to a mean of 50 (SD = 10) in the general U.S. population, where higher scores reflect better mental well-being. The change in SF-36 MCS scores was measured from baseline to 12 weeks.
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Game Intervention | No Intervention
Number analyzed (Participants) | 12 | 12
score on a scale | -0.3 (5.68) | 0.3 (9.18)
Statistical Analysis 1: Comparison: Game Intervention vs No Intervention; Null hypothesis: no improvement or worse with intervention Alternative hypothesis: improvement with intervention; Test type: Superiority; p = 0.432, t-test, 1 sided; The threshold for statistical significance was p=0.05

7. Secondary Outcome: Change in Lawton-Brody Instrumental Activities of Daily Living Scale (IADL)
Description: IADL scores range between 0 and 8. Higher scores indicate greater levels of performance in activities of daily living. The change in IADL scores was measured from baseline to 12 weeks
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Game Intervention | No Intervention
Number analyzed (Participants) | 12 | 12
score on a scale | -0.5 (1.66) | -0.1 (1.04)
Statistical Analysis 1: Comparison: Game Intervention vs No Intervention; Test type: Superiority — Null hypothesis: no improvement or worse with intervention Alternative hypothesis: improvement with intervention; p = 0.750, t-test, 1 sided

ADVERSE EVENTS:
Time Frame: 24 weeks
Description: daily questionnaire
Arm/Group | Game Intervention | No Intervention | Caregivers
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/12 | 0/2
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/12 | 0/2
Other Adverse Events (participants affected / at risk) | 0/12 | 0/12 | 0/2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2025-02-05): https://cdn.clinicaltrials.gov/large-docs/23/NCT04920123/Prot_000.pdf
  • Statistical Analysis Plan (2025-03-31): https://cdn.clinicaltrials.gov/large-docs/23/NCT04920123/SAP_001.pdf
  • Informed Consent Form (2023-10-06): https://cdn.clinicaltrials.gov/large-docs/23/NCT04920123/ICF_002.pdf